CLINICAL TRIAL: NCT04421443
Title: Feasibility and Clinical Usefulness of the Unified Protocol in Online Group Format for Bariatric Surgery Candidates: Study Protocol for a Multiple Baseline Experimental Design
Brief Title: Unified Protocol for Bariatric Surgery Candidates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jorge Javier Osma López (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Universidad de Zaragoza (Other)
Responsible Party: Sponsor-Investigator, Jorge Javier Osma López, Principal Investigator, Instituto de Investigación Sanitaria Aragón
Organization: Instituto de Investigación Sanitaria Aragón (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPES/CB/2020
Record Dates: First submitted 2020-05-26; First posted 2020-06-09 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Emotional Disorder; Anxiety; Depression
Keywords: Emotional Disorders; Transdiagnostic; Unified Protocol; Bariatric Surgery; Obesity; Emotional Regulation
MeSH Terms: conditions — Anxiety Disorders; Depression; Obesity; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: In the present investigation, all consecutive patients who have been selected to undergo bariatric surgery and present anxiety or depressive symptoms or at least one diagnosis of emotional disorder, are asked to participate. Once inclusion criteria are accomplished, each patient will be randomly assigned to one of the multiple baseline groups: 3, 5 or 8 evaluation days before the intervention. The study includes eleven assessment points (baseline, pre-treatment, post-treatment and eight follow-ups, one every three months until two years after treatment completion).
Who Masked: Participant
Masking Description: Participants will know the baseline condition they have been assigned to: 3, 5 or 8 evaluation days before the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3 days before intervention (Active Comparator): Participants have to complete a pre-treatment assessment (baseline) for 3 days.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- 5 days before intervention (Active Comparator): Participants have to complete a pre-treatment assessment (baseline) for 5 days.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- 8 days before intervention (Active Comparator): Participants have to complete a pre-treatment assessment (baseline) for 8 days.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — This intervention focuses on a wide range of emotional psychopathology, allowing care for comorbid disorders and subclinical or unspecified symptoms, which reduces treatment times and costs, and improves response to treatment. The intervention will be carried out in an online-group format. For ethical reasons, if any of the patients feel uncomfortable during the study with the online-group format, will may leave the group and receive individual attention. The study plans follow-ups every three months until two years after post-treatment, all of them will be conducted online.

SUMMARY:
The present pilot study with a multiple baseline experimental desing will verify the feasibility and clinical utility of the Unified Protocol, applied in an online group format in a mental health setting of the Spanish national health system to patients waiting for bariatric surgery with diagnosis or symptoms of Emotional Disorders

DETAILED DESCRIPTION:
Obesity is currently becoming a serious global public health problem due to the high prevalence and the large increase in recent years. This condition is associated with different health problems, including physical and mental diseases. The presence of anxiety or depression disorders among candidates for bariatric surgery it is very high and predicts worse results. The present study aims to explore the feasibility and clinical usefulness of an online group format application of the Unified Protocol, a transdiagnostic emotion-based intervention for patients waiting for bariatric surgery with at least one emotional disorder diagnosis or emotional symptoms.

We will conduct a pilot study with a repeated single case experimental design (multiple baseline design) in a public mental health service. The sample will consist of 45 participants who will be randomized to three baseline conditions: 8, 12 or 15 evaluation days before the intervention. Depression and anxiety symptoms and diagnostic criteria will be the primary outcome measures. Secondary measures will include evaluation of affectivity, personality traits, general fit, quality of life, and different body image and eating outcomes. An analysis of treatment satisfaction will be also performed. Assessment points include baseline, pre-treatment, post-treatment, and follow-ups every three months until two years after post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being of a legal age
* Being a bariatric surgery candidate
* Presenting anxious or depressive symptomatology (subclinical symptoms with BDI-II and BAI) or meeting the criteria for at least one emotional disorder (anxiety, mood and related disorders) from the International Neuropsychiatric Interview (MINI)
* Speaking Spanish or Catalan fluently
* Committing to attend the sessions
* Understanding and accepting the contents of the informed consent, expressed by signing it
* Having Internet to fulfill the protocol assessments online, and (8) being agree to maintain the prescribed medication regimen (including dosage) during the evaluation period, if any, and during treatment

Exclusion Criteria:

* Having a severe condition that would require to be prioritized for treatment, so that an interaction between both interventions cannot be ruled out. These include a severe mental disorder (bipolar disorder, personality disorder, schizophrenia, or an organic mental disorder), suicide risk at the time of assessment, or substance use in the last three months (excluding cannabis, coffee, and/or nicotine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini International Neuropsychiatric Interview (MINI) | Only before of the treatment to check inclusion criteria, an average of 3 months
  This interview contains structured questions that evaluate major psychiatric disorders based on the Diagnostic and Statistical Manual of Mental Disorders
Beck Anxiety Inventory (BAI) | Only before of the treatment to check inclusion criteria, an average of 3 months
  The BAI is composed of 21 items that evaluate anxiety symptoms. Responses use a 4-point Likert scale ranging from 0 (Not at all) to 3 (Severely). The total score can range from 0 to 63. Higher scores are indicative of greater severity and functional impairment as a result of anxious symptoms.
Beck Depression Inventory (BDI-II) | Only before of the treatment to check inclusion criteria, an average of 3 months
  It consists of 21 items, each with four different statements that reflect an increase in the degree of depression. A score of 0 indicates the absence of depressive symptoms and 3 reflects the most severe levels of depression. The scale has a 0-to-63 range. Higher scores are indicative of greater severity and functional impairment as a result of depressive symptoms.
Overall Depression Severity and Impairment Scale (ODSIS) | Up to 24 months
  Consist of five items that evaluate the frequency and the intensity of depressive symptoms and their interference with the person's work or school life and social life. The total score range from 0 to 20 and responses use a 5-point Likert scale ranging from 0 to 4. Higher scores are indicative of greater severity and functional impairment as a result of depressive symptoms.
Overall Anxiety Severity and Impairment Scale (OASIS) | Up to 24 months
  Consist of five items that evaluate the frequency and the intensity of anxious symptoms and their interference with the person's work or school life and social life. The total score range from 0 to 20 and responses use a 5-point Likert scale ranging from 0 to 4. Higher scores are indicative of greater severity and functional impairment as a result of anxious symptoms.

SECONDARY OUTCOMES:
Positive and Negative Affect Scale (PANAS) | Up to 24 months
  It consists of 20 items that measure both positive and negative affect, 10 items for each dimension. Each item is rated on a 5-point Likert scale ranging from 1 (Not at all, very slightly) to 5 (Extremely). The higher the score in each of the dimensions, the greater the affect evaluated
NEO Five-Factor Inventory (NEO-FFI) | Up to 24 months
  This scale contains 60 items that provide a quick and overall measurement of the five major personality factors. The responses are rated on a 5-point Likert scale ranging from 0 (Strongly agree) to 4 (Strongly disagree). The higher the score in each of the dimensions, the higher the tendency toward that personality factor
Quality of Life Index (QLI) | Up to 24 months
  It contains 10 items that are rated on a 10-point Likert scale ranging from 1 (Poor) to 10 (Excellent). The higher the score, the higher the quality of life
Maladjustment Inventory (MI) | Up to 24 months
  This scale reflects the extent to which the person's current problems are affecting the different areas of their daily life, which are scored on a 6-point Likert scale ranging from 0 (not at all ) to 5 (Very severe). The higher the score, the greater the interference of current problems in the person's life
Difficulties in Emotion Regulation Scale (DERS) | Up to 24 months
  This scale includes 28 items rated on a 5-point Likert scale ranging from 1 (almost never/0-10% of the time) to 5 (almost always/90-100% of the time). The higher the total score, the higher the emotional dysregulation
EuroQol | Up to 24 months
  It is a generic instrument that will be use to measure health-related quality of life. Have 5 dimensions (mobility, personal care, daily activities, pain and anxiety/depression), and a general state of health perceived by means of a visual analog scale
Bulimic Investigatory Test Edinburgh (BITE) | Up to 24 months
  It is a self-report questionnaire used to evaluate the presence and severity of bulimic symptomatology, and cognitive and emotional signs and symptoms associated with binge eating. The total of score for all questions will give you a symptom score of 15 or above indicates that you have a lot of the thoughts and attitudes consistent with an eating disorder.
Body Shape Questionnaire (BSQ) | Up to 24 months
  It is a self-applied questionnaire which is used to evaluate fear of putting on weight, feelings of low self-esteem because of one's appearance, the desire to lose weight and body dissatisfaction. The scores are classified in 4 categories: not worried about body shape <81, slightly worried = 81-110, moderately worried = 111-140, extremely worried >140.
Emotional Eating Scale (EES) | Up to 24 months
  It is a 25-item self-report measure that assesses a person's tendency to cope with emotions through food. Each of the 25 items evaluates a different emotion through specific adjectives. The adjectives are valued in a 5-point Likert-type format that assesses the relationship between the emotion and the intensity of the desire to eat it causes. It is scored on a scale of 0 to 4: 0-I don't feel like eating; 4-I have a desire to eat very strong. Higher scores are indicative of a greater tendency to regulate emotions through diet.
Mensual Body Mass Index (BMI) | Up to 24 months
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres. For most adults, an ideal BMI is in the 18.5 to 24.9 range. If the BMI is for below 18.5 - is in the underweight range; between 18.5 and 24.9: you are in the healthy weight range; between 25 and 29.9 - you are in the overweight range; between 30 and 39.9 - you are in the obesity range.
Satisfaction with Treatment | Through study completion, an average of 3 months
  This ad hoc questionnaire assesses participants' opinion of the treatment received, to what extent it has helped participants adaptively regulate emotions, and which techniques have most influenced the regulation of their emotions. Higher scores on the questionnaire show greater satisfaction towards the treatment received.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Osma, Ph. D., Principal Investigator — Instituto de Investigación Sanitaria Aragón, Universidad de Zaragoza
Locations (1):
- Instituto de investigación sanitaria de Aragón, universidad de Zaragoza, Teruel, Spain

IPD SHARING:
Plan to Share IPD: Yes
Under request

REFERENCES:
- See also: IPES web (Investigation group) — https://ipes-group.com/